CLINICAL TRIAL: NCT02896114
Title: A Retrospective Study of Surgical Treatment of Congenital Pseudarthrosis of Tibia in China: a Muti-centre Study
Brief Title: A Retrospective Study of Surgical Treatment of Congenital Pseudarthrosis of Tibia in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Children's Hospital (Other Government)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan Women and Children's Medical Center (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Beijing Children's Hospital (Other); Dalian Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Kunming Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HN03
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Congenital Pseudarthrosis of Tibia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to evaluate the current methods of surgical treatment for Congenital Pseudarthrosis of tibia(CPT) in children and their results respectively.

DETAILED DESCRIPTION:
The study aims to evaluate the current surgical treatment and its result for Congenital Pseudarthrosis of tibia (CPT)in children in China. A retrospective study will be conducted with around 150 patients at 11 centers in China. This study will use available registry data from a defined time period of Jan 2006-Dec 2014. The treatment method will be recorded. The bone union rate and the refracture rate were calculated to evaluate the final result of several surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria consists of patients with congenital pseudarthrosis of Tibia who were surgical treated to obtain bone union.

Exclusion Criteria:

* Patients are complicated with mental, neurological disorders (such as hypoxic-ischemic encephalopathy, epilepsy and dementia) or significant barriers to growth.
* Patients with pseudarthrosis of tibia caused by trauma, tumor,infection, etc
* Children are complicated with dysfunction of liver and kidney , blood disorders, immune deficiency disease and ECG abnormalities.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with congenital pseudarthrosis of Tibia who were surgical treated to obtain bone union.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
whether the tibial has obtained union | 9 months post-operation
  Ohnishi criterion: Degree of union was evaluated by the findings on radiographs and classified into three grades( Ohnishi criterion): union, delayed union, and nonunion. Radiographic union was defined as possessing continuity of bone density between the fragments without obvious radiolucent zone between them and possessing cortex-bridging fragments with sufficient thickness and radiodensity on both anteroposterior and lateral radiographs. Delayed union was defined as a process of healing that was slow but was progressing. Nonunion was defined by the healing process that had completely ceased.

SECONDARY OUTCOMES:
clinical outcome measurement(Johnston clinical evaluation criterion) | 9 months post-operation，the last follow up
  Johnston clinical evaluation criterion of Congenital Pseudarthrosis of Tibia (CPT): The outcome was classified as grade 1 when there was unequivocal union with full weight-bearing function and maintenance of alignment requiring no additional surgical treatment; grade 2 when there was equivocal union with useful function, with the limb protected by a brace, and/or valgus or sagittal bowing for which additional surgery was required or anticipated; and grade 3 when there was persistent nonunion or refracture, requiring full-time external support for pain and/or instability.
Refracture of tibia | Time Frame: 1,2,3,4,5,6,7,8,9 years post-operation,the last follow-up
  The continuity of tibia cortex was disappeared in X ray.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Yao, Principal Investigator — Hunan Children's Hospital
Locations (1):
- Hunan Children's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohnishi I, Sato W, Matsuyama J, Yajima H, Haga N, Kamegaya M, Minami A, Sato M, Yoshino S, Oki T, Nakamura K. Treatment of congenital pseudarthrosis of the tibia: a multicenter study in Japan. J Pediatr Orthop. 2005 Mar-Apr;25(2):219-24. doi: 10.1097/01.bpo.0000151054.54732.0b. PMID 15718906
- [Background] Romanus B, Bollini G, Dungl P, Fixsen J, Grill F, Hefti F, Ippolito E, Tudisco C, Wientroub S. Free vascular fibular transfer in congenital pseudoarthrosis of the tibia: results of the EPOS multicenter study. European Paediatric Orthopaedic Society (EPOS). J Pediatr Orthop B. 2000 Apr;9(2):90-3. doi: 10.1097/01202412-200004000-00003. PMID 10868357
- [Background] Mathieu L, Vialle R, Thevenin-Lemoine C, Mary P, Damsin JP. Association of Ilizarov's technique and intramedullary rodding in the treatment of congenital pseudarthrosis of the tibia. J Child Orthop. 2008 Dec;2(6):449-55. doi: 10.1007/s11832-008-0139-4. Epub 2008 Oct 28. PMID 19308541